CLINICAL TRIAL: NCT02910193
Title: Alcohol Addiction: A Systems-oriented Approach; Functional Validation II: Neuroimaging x Genetics
Brief Title: Alcohol Addiction: A Systems-oriented Approach
Acronym: eMedAlcohol
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Principal Investigator, Andreas Heinz, Prof., MD, PhD, Charite University, Berlin, Germany
Other Study IDs: 01ZX1311E
Record Dates: First submitted 2016-02-22; First posted 2016-09-21 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Alcoholism
Keywords: alcoholism; genetics; functional MRI; structural MRI; first-degree relatives
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — EDTA and PAX blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- alcohol-dependent patients
- first-degree relatives: Parents, children, siblings of alcohol-dependent patients
- healthy control subjects

SUMMARY:
The goal of the multicenter subproject (SP) 10 of the eMED Alcohol Addiction Consortium - A Systems-Oriented Approach is to study neuroimaging x genetics predictions in an existing sample (NGFNplus) of tightly endophenotyped and genome-wide genotyped alcohol dependent subjects (N=240) and controls (N=240); (ii) to translate the results of neuroimaging and genetic analyses from an adolescent risk sample (IMAGEN) to adult disease (NGFNplus sample) by examining related MRI-paradigms tagging the same functional brain systems in both samples (e.g. reward system, inhibitory control system, emotion processing, working memory); (iii) to conduct a follow-up neuroimaging study on the NGFNplus sample validating the neurobehavioral risk profiles predictive for juvenile harmful alcohol use in adult patients with alcohol addiction, (iv) to expand the NGFNplus sample by including a new set of healthy subjects with high genetic risk (1st degree relatives of patients with alcohol addiction). The investigators will do so by using elaborate imaging genetic methods that are already available and successfully used in other multicenter studies by the investigator's research group (e.g. univariate analyses, functional and effective connectivity analyses, polygenetic scores, network topology) as well as by using complex computational algorithms and mathematical models, in particular advanced machine learning methods, developed in SP 6. The investigator's approach aims in the long to predict and characterize longitudinal outcomes in patients with alcohol addiction (5 years following our index session) and to complement the NGFN-sample with an add-on study with 1st degree relatives that will allow the investigators to test the generalizability of the identified predictive risk profiles for early risk identification.

DETAILED DESCRIPTION:
The overall research goal of this project is (i) to study neuroimaging x genetics predictions in an existing sample (NGFNplus) of tightly endophenotyped and genome-wide genotyped alcohol dependent subjects (N=240) and controls (N=240); (ii) to translate the results of neuroimaging x genetic analyses from an adolescent risk sample (IMAGEN) to adult disease (NGFNplus sample) by examining related paradigms tagging the same functional systems in both samples; (iii) to conduct a follow-up neuroimaging study on the NGFNplus sample validating the neurobehavioral risk profiles predictive for harmful alcohol use in adolescents in adult patients with alcohol addiction (iv) to expand the NGFNplus sample by including a new set of healthy subjects with high genetic risk (1st degree relatives of patients with alcohol addiction). The investigators will do so by using imaging genetic methods that are already available and used in other multicenter studies by the investigator's research group (e.g. univariate analyses, functional and effective connectivity analyses, polygenetic scores, network topology) as well as by using computational algorithms and mathematical models, in particular advanced machine learning methods, developed in other sub projects (SPs) of the consortium in particular of SP4 and SP6. The investigator's approach will enable the researchers to characterize outcome longitudinal in patients with alcohol addiction (5 years following our index session) and to complement the NGFN-sample with an add-on study with 1st degree relatives that will allow the investigators to test the generalizability of the identified predictive risk profiles for early risk identification.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* right handedness
* no psychiatric disorders according to the International Classification of Diseases, Version 10 (ICD-10) (in patients: other than nicotine and alcohol dependence)
* no use of psychotropic substances during previous 3 months

Exclusion Criteria:

* severe illnesses (e.g. neurological diseases)
* MR-contraindications (e.g. pacemaker, metal or electronic implants, metal splinters)
* no psychiatric axis I-disorders according to the International Classification of Diseases, Version 10 (ICD-10) (in patients: other than nicotine and alcohol dependence)
* no use of psychotropic substances during previous 3 months
* insufficient language knowledge
* claustrophobia
* pregnancy in women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic and community sample
Sampling Method: Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2016-05-17 (Actual); Primary Completion 2019-05-27 (Actual); Study Completion 2019-05-27 (Actual)

PRIMARY OUTCOMES:
Functional brain imaging assessed using a Siemens Magnetom TimTrio, 3 Tesla | 3 year
  The primary outcome measure "Blood Oxygenation Level-Dependent (BOLD) response" will be assessed as a marker of neural activation via functional brain imaging (fMRI) during the processing of emotional, monetary and alcohol-associated cues as well as cognitive demand and at rest. A Siemens Magnetom TimTrio, 3 Tesla will be used.
Structural brain imaging assessed using a Siemens Magnetom TimTrio, 3 Tesla | 3 year
  The second primary outcome measure "brain tissue (Grey Matter, White Matter, Cerebrospinal fluid)" will be assessed and quantified via structural brain imaging using magnet resonance tomography as well as defusion-tensor imaging (MRI, DTI). A Siemens Magnetom TimTrio, 3 Tesla will be used.

SECONDARY OUTCOMES:
Assessment of genetic candidate markers and epigenetic markers of alcohol use disorders | 3 years
  Secondary outcome measures will be genotype specification of candidate SNPs (e.g. BDNF, GATA4, OPRM1, D2/D1) derived from blood samples and according DNA/RNA array genotyping. Project aim is to conduct Genom-Wide Association Studies (GWAS) to investigate genetic factors that may predispose to or protect against alcohol use disorder. Further epigenetic methylation factors (i.e. homocysteine serum level) will be investigated to differentiate between healthy controls, alcohol-dependent patients and individuals at risk (first grade relatives).

CONTACTS AND LOCATIONS:
Locations (1):
- Charite - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared within the study consortium "SysMedAlcoholism".

REFERENCES:
- [Background] Spanagel R, Durstewitz D, Hansson A, Heinz A, Kiefer F, Kohr G, Matthaus F, Nothen MM, Noori HR, Obermayer K, Rietschel M, Schloss P, Scholz H, Schumann G, Smolka M, Sommer W, Vengeliene V, Walter H, Wurst W, Zimmermann US; Addiction GWAS Resource Group; Stringer S, Smits Y, Derks EM. A systems medicine research approach for studying alcohol addiction. Addict Biol. 2013 Nov;18(6):883-96. doi: 10.1111/adb.12109. PMID 24283978
- See also: Related Info — http://www.sys-med.de/en/consortia/sysmedalcoholism/